CLINICAL TRIAL: NCT01808560
Title: Pilot Study for Treatment of Meibomian Gland Dysfunction (MGD) Prior to Cataract Surgery
Brief Title: Treatment of Meibomian Gland Dysfunction Prior to Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TearScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LF005
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Blepharitis; Dry Eye Syndrome
MeSH Terms: conditions — Blepharitis; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LipiFlow Pre-treatment (Experimental): Subjects randomized to the LipiFlow Pre-Treatment group receive a 12-minute LipiFlow System treatment for MGD in both eyes one month prior to cataract surgery.
  Interventions: Device: LipiFlow Pre-Treatment
- Untreated Control (No Intervention): Subjects randomized to the untreated control group receive no MGD treatment prior to cataract surgery.
- LipiFlow Post-treatment (Experimental): Subjects in the untreated control group receive a 12-minute crossover treatment with the LipiFlow System in both eyes three months after cataract surgery.
  Interventions: Device: LipiFlow Post-treatment

INTERVENTIONS:
Device: LipiFlow Pre-Treatment — The LipiFlow Thermal Pulsation System is intended for the application of localized heat and pressure therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction, also known as evaporative dry eye or lipid deficiency dry eye.
  Other Names: LipiFlow Thermal Pulsation System
  Arms: LipiFlow Pre-treatment
Device: LipiFlow Post-treatment — The LipiFlow Thermal Pulsation System is intended for the application of localized heat and pressure therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction, also known as evaporative dry eye or lipid deficiency dry eye.
  Other Names: LipiFlow Thermal Pulsation System
  Arms: LipiFlow Post-treatment

SUMMARY:
The purpose of this pilot feasibility study is to assess whether treating meibomian gland dysfunction (MGD) prior to cataract surgery helps promote meibomian gland function, visual quality and ocular comfort after cataract surgery.

DETAILED DESCRIPTION:
This is a post-market, prospective, non-significant risk, open-label, randomized multi-center clinical trial evaluating treatment with the LipiFlow System in patients with meibomian gland dysfunction prior to planned bilateral cataract surgery. All subjects undergo examination to determine study eligibility and to capture the Baseline status prior to surgery. Subjects are randomized to receive LipiFlow treatment (Pre-treatment group) one month before cataract surgery or no LipiFlow treatment (Untreated Control group). Cataract surgery is performed on both eyes of each subject with the second eye surgery completed within two months of the first eye. All subjects are evaluated at one month and three months after cataract surgery on the second eye with comparison of the study endpoints between the Pre-treatment and Untreated groups. To facilitate subject recruitment, the Untreated Control group receives crossover LipiFlow treatment for MGD (Post-treatment group) three months after cataract surgery on the second eye.

ELIGIBILITY:
Inclusion Criteria:

* 55 to 85 years of age
* Must be able to comply with protocol including study randomization; completion of planned bilateral cataract surgery; no use of other MGD or dry eye treatments during the study; and attendance at all study visits
* Meibomian gland dysfunction in both eyes based on total meibomian gland score
* None to mild dry eye symptoms based on Ocular Surface Disease Index score
* Tear film interferometry assessment of 100 units or less

Exclusion Criteria:

* Systemic disease conditions that causes dry eye
* Use of systemic medications known to cause dry eye
* Use of other MGD or dry eye treatments except for over the counter lubricants or dietary supplements
* History of any of the following ocular conditions in the past 3 months: surgery, trauma, Herpes infection, recurrent inflammation, punctal plug insertion or punctal occlusion
* Presence of any of the following active conditions: ocular infection, ocular inflammation, moderate to severe allergic conjunctivitis, severe eyelid inflammation, eyelid abnormality that affects lid function, or ocular surface abnormality that compromises corneal integrity
* Participation in another ophthalmic drug or device trial in the past month

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Stevens, OD, MPH, Study Director — TearScience
Locations (7):
- United States (7):
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois
  - Jackson Eye, Lake Villa, Illinois
  - Charles River Eye Associates, Winchester, Massachusetts
  - Associated Eye Care, Stillwater, Minnesota
  - Ophthalmology Consultants, Ltd., St Louis, Missouri
  - The May Eye Care Center, Hanover, Pennsylvania
  - Carolina EyeCare Physicians, LLC, Mt. Pleasant, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Randomization and Treatment Allocation
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Started | 18 | 16 | 0
Completed | 18 | 16 | 0
Not Completed | 0 | 0 | 0
Period: 1-Month After Cataract Surgery
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Started | 16 (ITT: 2 subjects withdrew b/c they were unable to complete cataract surgery scheduled for both eyes) | 13 (ITT: 3 subjects withdrew b/c they were unable to complete cataract surgery scheduled for both eyes) | 0
Completed | 16 | 13 | 0
Not Completed | 0 | 0 | 0
Period: 3-Month After Cataract Surgery
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Started | 17 | 13 | 0
Completed | 17 | 13 | 0
Not Completed | 0 | 0 | 0
Period: Crossover Treatment
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Started | 0 | 0 | 13 (Post-Treatment Group Received Crossover LipiFlow treatment 3 Months after cataract surgery)
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 0
Period: 4-Month After Cataract Surgery
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Started | 0 | 0 | 13
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment | Total
Number analyzed (Participants) | 18 | 16 | 0 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (5.7) | 68.6 (6.4) |  | 70.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 |  | 25
  Male | 5 | 4 |  | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  | 1
  Not Hispanic or Latino | 17 | 16 |  | 33
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 |  | 1
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 1 | 0 |  | 1
  White | 17 | 15 |  | 32
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Total Meibomian Gland Score
Description: The primary endpoint is the mean change in total meibomian gland score in the Pre-treatment group compared to the Untreated group from Baseline after cataract surgery.
  Meibomian gland assessment was performed to evaluate the function of the meibomian glands based on the secretion characteristics from the gland orifices along the lower eyelid. Under a slit-lamp biomicrosope, the gland orifices were evaluated using a handheld instrument, Meibomian Gland Evaluator. This instrument provided a standardized method of applying the same amount of pressure and for each eye to ensure measurement consistency. A total of 15 glands were evaluated including five glands each in the temporal, central and nasal regions of the lower eyelid. For each gland, secretion characteristics were graded as 3 (clear liquid), 2 (cloudy liquid), 1 (inspissated/toothpaste consistency) and 0 (no secretion). The total meibomian gland score is the sum of the grades for all 15 glands with a range of 0 to 45.
Time Frame: Baseline and 3 Months post-surgery
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (Standard Deviation); unit: Change in Meibomian Gland Score
Units Other Than Participants: Eyes
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Number analyzed (Participants) | 17 | 13 | 0
Number analyzed (Eyes) | 34 | 26 | 0
Change in Meibomian Gland Score | 12.8 (9.9) | 1.9 (6.1) |

2. Secondary Outcome: Mean Change in Dry Eye Questionnaire Score From Baseline at 3 Months
Description: Assess for reduction in dry eye symptoms in symptomatic contact lens after LipiFlow treatment in comparison to an untreated control using Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire. It was defined as the mean change in SPEED score in the LF Treatment group compared to Control group from Baseline to 3 Months. The symptoms assessed are dryness, grittiness / scratchiness; soreness / irritation; burning / watering; and eye fatigue. Symptom frequency is on a scale of: 0 (never), 1(sometimes), 2 (often) and 3 (constant). Symptom severity is on a scale of: 0 (no problems), 1 (tolerable-not perfect but not uncomfortable), 2 (uncomfortable-irritating but does not interfere with my day), 3 (bothersome-irritating and interferes with my day) and 4 (intolerable-unable to perform my daily tasks). SPEED score is calculated as sum of frequency and severity scores for symptoms over a range from 0 to 28. A lower SPEED score represents less frequent and/or less severe symptoms.
Time Frame: Baseline and 3 Months post-surgery
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (Standard Deviation); unit: Change in SPEED Score
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Number analyzed (Participants) | 17 | 13 | 0
Change in SPEED Score | -3.4 (5.7) | 1.2 (5.4) |

3. Other Pre Specified Outcome: Mean Change in Ocular Surface Disease Index (OSDI) Questionnaire Score From Baseline at 3 Months
Description: Dry eye symptoms assessed using the OSDI questionnaire are sensitivity to light, grittiness, pain or soreness, blurred vision and poor vision. The assessment considers the frequency that problems with the eyes limit performance in reading, driving at night, working with a computer or bank machine, and watching television. Also, the frequency that eyes feel uncomfortable is assessed in windy conditions, areas with low humidity, and air-conditioned areas. The frequency scale is: 0 (none of the time), 1 (some of the time), 2 (half of the time), 3 (most of the time) and 4 (all of the time). The subject can answer not applicable (N/A) if the subject did not experience the situation or condition in the past week. Total OSDI score is calculated as the sum of frequency scores for all symptoms multiplied by 25 and divided by the number of questions answered with a range from 0 to 100. A lower OSDI score represents less disability from dry eye symptoms.
Time Frame: Baseline and 3 Months post-surgery
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (Standard Deviation); unit: Change in Total OSDI Score
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Number analyzed (Participants) | 17 | 13 | 0
Change in Total OSDI Score | -8.7 (22.3) | 2.0 (17.2) |

4. Other Pre Specified Outcome: Mean Change in NEI-VFQ Questionnaire Score From Baseline at 3 Months
Description: The National Eye Institute Visual Function Questionnaire (NEI-VFQ) evaluates frequency or severity of a symptoms and the effect on activities of daily living.
  The questionnaire has an overall score and 12 subscale scores for general health, general vision, ocular pain, difficulty with near vision activities, difficulty with distance vision activities, social functioning limitations due to vision, mental functioning limitations due to vision, role limitations due to vision, dependency on others due to vision, driving difficulties, color vision and peripheral vision.
  The NEI-VFQ scores range from 0 to 100 with lower scores indicating more symptoms or difficulty with activities of daily living. The questionnaire is scored by recoding responses to set values on a 0 to 100 scale such that the lowest value is set to 0 and the highest value is set to 100. The overall score is the average of vision subscale scores, excluding general health question.
Time Frame: Baseline and 3 Months post-surgery
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (Standard Deviation); unit: Change in NEI-VFQ-25 Composite Score
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Number analyzed (Participants) | 17 | 13 | 0
Change in NEI-VFQ-25 Composite Score | 11.6 (14.1) | 7.3 (10.8) |

5. Other Pre Specified Outcome: Mean Change in Number of MGYLS (Meibomian Glands Yielding Liquid Secretion)
Description: Meibomian gland assessment was performed to evaluate the function of the meibomian glands based on the secretion characteristics from the gland orifices along the lower eyelid at the visits. Under a slit-lamp biomicrosope, the gland orifices were evaluated using a handheld instrument, Meibomian Gland Evaluator, to apply gentle pressure along the eyelid margin. This instrument provided a standardized method of applying the same amount of pressure at each visit and for each eye to ensure measurement consistency.
  The number of meibomian glands yielding liquid secretion (MGYLS) (i.e., cloudy or clear liquid with a grade of 2 or 3) was counted out of the 15 glands assessed with a range of 0 to 15. A higher total meibomian gland score or higher number of MGYLS reflects less meibomian gland dysfunction.
Time Frame: Baseline and 3 Months post-surgery
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (Standard Deviation); unit: Change in Number of MGYLS
Units Other Than Participants: Eyes
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Number analyzed (Participants) | 17 | 13 | 0
Number analyzed (Eyes) | 34 | 26 | 0
Change in Number of MGYLS | 5.6 (4.8) | 1.0 (3.1) |

6. Other Pre Specified Outcome: Mean Change in Tear Break-up Time (TBUT)
Description: The Investigator or designee measures tear break-up time (TBUT) under a slit-lamp biomicroscope following instillation of fluorescein dye in the eye using the Dry Eye Test (DET) method.
  Tear film break-up is defined as the first observed break-up of the tear film following the third blink. Using a stopwatch to record the time, start the stopwatch as soon as the subject opens his/her eyes after the third blink and stop the stopwatch when the first break-up of the tear film is observed.
  Any values recorded as greater than 20 seconds were converted to 20 seconds in the analysis. Three separate measurements were taken for each eye and were averaged for analysis. A higher tear break-up time indicates better tear film stability.
Time Frame: Baseline and 3 Months post-surgery
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (Standard Deviation); unit: Change in TBUT (in seconds)
Units Other Than Participants: Eyes
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
Number analyzed (Participants) | 17 | 13 | 0
Number analyzed (Eyes) | 34 | 26 | 0
Change in TBUT (in seconds) | 1.4 (5.2) | -0.6 (3.0) |

ADVERSE EVENTS:
Arm/Group | LipiFlow Pre-treatment | Untreated Control | LipiFlow Post-treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 18 months of Sponsor's receipt of data from all sites, Investigators may publish or present the Investigator's individual results. Investigator must submit materials to Sponsor for review and comment at least 30 days prior to presentation or submission for publication. Investigator will consider all reasonable comments from Sponsor. Upon Sponsor's written request, Investigator agrees to delete any Proprietary Information other than Investigator's individual Study results.